CLINICAL TRIAL: NCT02239224
Title: A Placebo-Controlled, Randomized, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK), and Biological Activity of ATYR1940 in Adult Patients With Molecularly Defined Genetic Muscular Dystrophies
Brief Title: Safety, Tolerability, Pharmacokinetics, and Biological Activity of ATYR1940 in Adult Participants With Muscular Dystrophy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: aTyr Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATYR1940-C-002; 2014-001753-17 (EudraCT Number)
Record Dates: First submitted 2014-09-07; First posted 2014-09-12 (Estimated); Results first posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-07

CONDITIONS: Facioscapulohumeral Muscular Dystrophy (FSHD)
Keywords: FSHD
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1: ATYR1940 0.3 mg/kg (Experimental): Participants will receive ATYR1940 0.3 milligrams/kilograms (mg/kg) intravenous (IV) infusion once weekly for 4 weeks.
  Interventions: Biological: ATYR1940
- Cohort 2: ATYR1940 1.0 mg/kg (Experimental): Participants will receive ATYR1940 1.0 mg/kg IV infusion once weekly for 4 weeks.
  Interventions: Biological: ATYR1940
- Cohort 3: ATYR1940 3.0 mg/kg (Experimental): Participants will receive ATYR1940 3.0 mg/kg IV infusion once weekly for 12 weeks.
  Interventions: Biological: ATYR1940
- Placebo (Placebo Comparator): Participants will receive placebo matched to ATYR1940 IV infusion once weekly for 4 weeks in Cohorts 1 and 2 and for 12 weeks in Cohort 3.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Placebo — Concentrate for solution for infusion
  Arms: Placebo
Biological: ATYR1940 — Concentrate for solution for infusion
  Arms: Cohort 1: ATYR1940 0.3 mg/kg; Cohort 2: ATYR1940 1.0 mg/kg; Cohort 3: ATYR1940 3.0 mg/kg

SUMMARY:
The purpose of this study is to assess the safety and tolerability profile of ATYR1940 in the treatment of adult participants with molecularly defined genetic muscular dystrophies

DETAILED DESCRIPTION:
Study ATYR1940-C-002 is a multi-national, multi-center, double-blind, randomized, placebo-controlled, ascending dose study designed to evaluate the safety, tolerability, PK, immunogenicity, and pharmacodynamic effects of ATYR1940 in participants with FSHD. Up to 44 participants are planned to be enrolled at multiple study centers in the United States and Europe; the actual number of participants enrolled will depend on the number of cohorts initiated.

Participants will be screened for study eligibility during the Screening period within 3 weeks before Baseline (that is, Day 1, the first day of Study Drug administration). Eligible participants, based on Screening assessments, will be randomly assigned to treatment with ATYR1940 or placebo. Participants who are randomized will be considered enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a male or female aged 18 to 65 years, inclusive.
* Participant has an established, genetically-confirmed, diagnosis of FSHD with clinical findings meeting existing criteria.
* Participant has provided written informed consent after the nature of the study has been explained and prior to the performance of any research-related procedures.
* Participant is, in the Investigator's opinion, willing and able to comply with all study procedures.
* Cohorts ≥2 only: Participant has imaging findings meeting defined criteria for muscle inflammation in at least 1 skeletal muscle.

Exclusion Criteria:

* Participant is currently receiving treatment with an immunomodulatory agent or has a history of such treatment, including targeted biological therapies (for example, etanercept, omalizumab) within the 3 months before Baseline; corticosteroids within 4 weeks before Baseline; or high-dose non-steroidal anti-inflammatory agents (NSAIDs) within 2 weeks before Baseline.
* Participant is currently receiving curcumin or albuterol or requires such treatment during study participation.
* Participant has evidence of an alternative diagnosis other than FSHD, based on prior muscle biopsy or genetic test findings.
* Participant has a presumptive diagnosis of FSHD, based on clinical assessment, but does not yet have genetic confirmation of the diagnosis.
* Participant has a severe retinopathy.
* Participant has a history of obstructive or restrictive lung disease (including interstitial lung disease, pulmonary fibrosis, or asthma), or evidence for interstitial lung disease on Screening chest radiograph.
* Participant has a history of anti-synthetase syndrome, prior Jo-1 antibody (Ab)-positivity, or has a positive or equivocally positive Jo-1 Ab test result during Screening.
* Participant has acute or clinically relevant Epstein-Barr virus or cytomegalovirus infection or re-activation.
* Participant has a chronic infection such as hepatitis B virus, hepatitis C virus, or human immunodeficiency virus or a history of tuberculosis.
* Participant has received a vaccination within 8 weeks before Baseline or vaccination is planned during study participation.
* Participant has symptomatic cardiomyopathy or severe cardiac arrhythmia that may, in the Investigator's opinion, limit the participant's ability to complete the study protocol.
* Participant has anemia (as defined for participant's age and gender by local laboratory range).
* Participant has gamma-glutamyl transferase (GGT) or serum creatinine levels >2 × the upper limit of normal (ULN).
* Participant has abnormal baseline findings, medical condition(s), or laboratory findings that, in the Investigator's opinion, might jeopardize participant's safety or decrease the chance of obtaining satisfactory data needed to achieve the objectives of the study.
* Participant has evidence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematological, metabolic, dermatological, or gastrointestinal disease, or has a condition that requires immediate surgical intervention or other treatment or may not allow safe participation.
* Participant has used any investigational product or device (other than a mobility assistance device) within 30 days before Baseline.
* Participant has received a product intended to enhance muscle growth within 30 days before Baseline.
* Participant underwent muscle biopsy within 30 days before Baseline.
* Participant initiated treatment with a statin or had a significant adjustment to their statin regimen within 3 months before Baseline. (Stable, chronic statin use is permissible.)
* Participant has received a product that putatively enhances muscle growth (for example, insulin-like growth factor, growth hormone) or activity (for example, Coenzyme A) on a chronic basis within 4 weeks before Baseline.
* Participant is unwilling to abstain from strenuous physical activity for 24 hours prior to each study center visit.
* Participant previously received ATYR1940.
* If female and of childbearing potential (premenopausal and not surgically sterile), participant has a positive pregnancy test at Screening or is unwilling to use contraception from the time of Screening through 1 month after the last Study Drug dose. Acceptable methods of birth control include abstinence, barrier methods, hormones, or intra-uterine device.
* If male, participant is unwilling to use a condom plus spermicide during sexual intercourse from the time of Screening through 1 month after the last Study Drug dose.
* Cohorts ≥2 only: Participant has a known contraindication for magnetic resonance imaging (MRI) assessments (for example metal prosthesis or pacemaker) as per local site MRI protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09-04 (Actual); Primary Completion 2015-12-14 (Actual); Study Completion 2015-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Shukla, MD, Study Director — aTyr Pharma
Locations (5):
- United States (2):
  - aTyr Pharma Investigative Site, Rochester, New York
  - aTyr Pharma Investigative Site, Columbus, Ohio
- aTyr Pharma Investigative Site, Marseille, France
- aTyr Pharma Investigative Site, Rome, Italy
- aTyr Pharma Investigative Site, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: ATYR1940 0.3 mg/kg: Participants received ATYR1940 0.3 milligrams/kilograms (mg/kg) intravenous (IV) infusion once weekly for 4 weeks.
- Cohort 2: ATYR1940 1.0 mg/kg: Participants received ATYR1940 1.0 mg/kg IV infusion once weekly for 4 weeks.
- Cohort 3: ATYR1940 3.0 mg/kg: Participants received ATYR1940 3.0 mg/kg IV infusion once weekly for 12 weeks.
- Placebo: Participants received placebo matched to ATYR1940 IV infusion once weekly for 4 weeks in Cohorts 1 and 2 and for 12 weeks in Cohort 3.
Period: Overall Study
Arm/Group | Cohort 1: ATYR1940 0.3 mg/kg | Cohort 2: ATYR1940 1.0 mg/kg | Cohort 3: ATYR1940 3.0 mg/kg | Placebo
Started | 3 | 6 | 6 | 5
Received at Least One Dose of Study Drug | 3 | 6 | 6 | 5
Completed | 3 | 6 | 3 | 4
Not Completed | 0 | 0 | 3 | 1
Not completed — Administrative | 0 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) analysis set included all participants who were randomized and received at least 1 dose (full or partial) of study drug.
Groups:
- Cohort 1: ATYR1940 0.3 mg/kg: Participants received ATYR1940 0.3 mg/kg IV infusion once weekly for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: ATYR1940 0.3 mg/kg | Cohort 2: ATYR1940 1.0 mg/kg | Cohort 3: ATYR1940 3.0 mg/kg | Placebo | Total
Number analyzed (Participants) | 3 | 6 | 6 | 5 | 20
Age, Continuous [Mean (Full Range); unit: years] | 44.3 [25 to 55] | 44.5 [33 to 52] | 45.3 [25 to 72] | 54.0 [39 to 66] | 49.35 [25 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 2 | 1 | 8
  Male | 2 | 2 | 4 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as adverse events (AEs) with an onset following administration of the first dose of study drug. An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with study drug. Worsening of a pre-existing medical condition, (that is, diabetes, migraine headaches, gout) should have been considered an AE if there was either an increase in severity, frequency, or duration of the condition or an association with significantly worse outcomes. Classification of AEs was to be done by the Investigator according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (up to Week 25)
Population: ITT analysis set included all participants who were randomized and received at least 1 dose (full or partial) of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ATYR1940 0.3 mg/kg | Cohort 2: ATYR1940 1.0 mg/kg | Cohort 3: ATYR1940 3.0 mg/kg | Placebo
Number analyzed (Participants) | 3 | 6 | 6 | 5
Participants | 3 | 6 | 6 | 5

2. Primary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA)
Description: Titers through Week 14 are summarized. For Cohorts 1 and 2, samples that screened positive but did not confirm on confirmatory assay were not titered.
Time Frame: Baseline up to Week 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ATYR1940 0.3 mg/kg | Cohort 2: ATYR1940 1.0 mg/kg | Cohort 3: ATYR1940 3.0 mg/kg | Placebo
Number analyzed (Participants) | 3 | 6 | 6 | 5
Participants | 2 | 1 | 3 | 0

3. Primary Outcome: Number of Participants With a Positive or Equivocal Jo-1 Antibody (Ab) Test Result
Description: Criterion for a positive Jo-1 Ab test result: >10.0 units/milliliter (U/mL), a cut-point associated with anti-synthetase syndrome. Criterion for an equivocal Jo-1 Ab test result: 7.0 to 10.0 U/mL. Participants were required to have a negative Jo-1 Ab test result (defined as <7 U/mL) for inclusion in the study as well as to continue dosing with study drug during the study.
Time Frame: Baseline up to Week 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ATYR1940 0.3 mg/kg | Cohort 2: ATYR1940 1.0 mg/kg | Cohort 3: ATYR1940 3.0 mg/kg | Placebo
Number analyzed (Participants) | 3 | 6 | 6 | 5
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With a Clinically Significant Laboratory Abnormality
Description: Laboratory parameters included hematology (hematocrit, hemoglobin, platelet count, red blood cell count, white blood cell count, neutrophils, lymphocytes, monocytes, eosinophils, basophils); serum chemistries (blood urea nitrogen, creatinine, total bilirubin, aspartate aminotransferase, alanine aminotransferase, gamma-glutamyl transferase (GGT), alkaline phosphatase, sodium, total protein, bicarbonate, potassium, calcium, chloride, magnesium, inorganic phosphate, creatine phosphokinase [will be fractionated if elevated], lactic dehydrogenase, erythrocyte sedimentation rate, C-reactive protein, troponin, myoglobin, insulin-like growth factor 1, cholesterol [non-fasting]); Urinalysis (Color, pH, specific gravity, protein, glucose, ketones, blood). Clinically significant laboratory abnormalities were based upon Investigator's discretion. A summary of all Serious AEs and Other AEs (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Baseline up to Week 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ATYR1940 0.3 mg/kg | Cohort 2: ATYR1940 1.0 mg/kg | Cohort 3: ATYR1940 3.0 mg/kg | Placebo
Number analyzed (Participants) | 3 | 6 | 6 | 5
Participants | 0 | 2 | 0 | 0

5. Primary Outcome: Number of Participants With a Physical Examination Abnormality
Description: Body systems that were evaluated during the physical examination included general appearance, head, eyes, ears, nose, throat (HEENT), cardiovascular system, respiratory system, chest (breasts), gastrointestinal system (abdomen), lymphatic system, musculoskeletal system, skin, psychiatric, and neurologic. Neurologic examination included assessment of mental status, memory, cranial nerves, motor function, and reflexes, and sensory testing. The body systems with at least 1 physical abnormality is presented. One participant could be represented in more than 1 body system category. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (up to Week 25)
Population: ITT analysis set included all participants who were randomized and received at least 1 dose (full or partial) of study drug. Here, 'Overall Number of Participants Analyzed' (N) signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ATYR1940 0.3 mg/kg | Cohort 2: ATYR1940 1.0 mg/kg | Cohort 3: ATYR1940 3.0 mg/kg | Placebo
Number analyzed (Participants) | 3 | 4 | 3 | 4
Participants
  General appearance | 0 | 1 | 0 | 0
  HEENT | 0 | 1 | 0 | 0
  Lymphatic system | 0 | 0 | 0 | 1
  Musculoskeletal system | 0 | 1 | 0 | 1
  Respiratory system | 0 | 1 | 0 | 0
  Skin | 0 | 1 | 1 | 0

6. Primary Outcome: Number of Participants With a Vital Sign-Related Event Resulting in a TEAE
Description: The vital sign parameters that were evaluated included heart rate, systolic and diastolic blood pressure, and respiration rate as well as temperature. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (Up to Week 25)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ATYR1940 0.3 mg/kg | Cohort 2: ATYR1940 1.0 mg/kg | Cohort 3: ATYR1940 3.0 mg/kg | Placebo
Number analyzed (Participants) | 3 | 6 | 6 | 5
Participants | 0 | 0 | 1 | 0

7. Primary Outcome: Number of Participants With a Pulmonary Function Event Resulting in a TEAE
Description: Pulmonary function testing included measurements of forced vital capacity (FVC) and forced expiratory volume in 1 second (FEV1). A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Up to End of Study (Up to Week 25)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ATYR1940 0.3 mg/kg | Cohort 2: ATYR1940 1.0 mg/kg | Cohort 3: ATYR1940 3.0 mg/kg | Placebo
Number analyzed (Participants) | 3 | 6 | 6 | 5
Participants | 0 | 1 | 0 | 0

8. Secondary Outcome: Percent Change From Baseline in Manual Muscle Testing (MMT) Score at Week 6 and Week 14
Description: MMT was graded on a scale from 0 (no movement) to 10 (normal movement). Each side of the body and the position in which each muscle was tested were recorded for each participant. The total MMT score were calculated by averaging a converted MMT scores across all tested muscle groups. Decreased motor function was indicated by decreased individual muscle or composite MMT score.
Time Frame: Baseline, Week 6 and Week 14
Population: ITT analysis set included all participants who were randomized and received at least 1 dose (full or partial) of study drug. Here, 'Number Analyzed' signifies participants evaluable at specified timepoints.
Measure: Mean (Full Range); unit: percent change
Arm/Group | Cohort 1: ATYR1940 0.3 mg/kg | Cohort 2: ATYR1940 1.0 mg/kg | Cohort 3: ATYR1940 3.0 mg/kg | Placebo
Number analyzed (Participants) | 3 | 6 | 6 | 5
percent change
  Change at Week 6 | 2.83 [1.0 to 4.4] | 3.07 [0.7 to 5.6] | -0.85 [-5.1 to 5.5] | 1.34 [-3.3 to 7.8]
  Change at Week 14: number analyzed (Participants) | 0 | 0 | 6 | 2
  Change at Week 14 |  |  | 0.70 [-5.9 to 9.2] | -1.40 [-1.5 to -1.3]

9. Secondary Outcome: Change From Baseline in Individualized Neuromuscular Quality of Life (INQoL) - Overall QoL at Week 6 and Week 14
Description: The INQoL is a validated muscle disease-specific measure of quality of life. The self-administered questionnaire consisted of 45 questions with 4 domains measuring the impact of common muscle disease symptoms (weakness, locking [or myotonia], pain, and fatigue); 5 domains measuring the influence of the muscle disease on particular areas of life (activities, independence, relationships, emotions, and body image); and the last domain focused on the positive and negative effects of treatment and was divided into 2 scores. All responses were given in a 7-point Likert scale, with improved QoL indicated by decreased scores. Overall QoL score was calculated from preselected 5 domains (activities, independence, relationships, emotions, and body image) by adding the scores from each domain. In summary, INQoL yielded 11 scores and 1 QoL score. The Overall scoring used a scale of 0-100, with improved QoL indicated by decreased scores.
Time Frame: Baseline, Week 6 and Week 14
Population: Per-Protocol (PP) analysis set included all participants in the ITT analysis set with no major protocol deviations and ≥1 post-baseline pharmacodynamic (PD) or clinical parameter assessed. Change from baseline included only those participants with both a baseline value and a value for the summarized time period. Here, 'Number Analyzed' signifies participants evaluable at specified timepoints.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Cohort 1: ATYR1940 0.3 mg/kg | Cohort 2: ATYR1940 1.0 mg/kg | Cohort 3: ATYR1940 3.0 mg/kg | Placebo
Number analyzed (Participants) | 3 | 6 | 6 | 5
score on a scale
  Baseline | 54.37 [36.8 to 68.4] | 72.80 [63.2 to 84.2] | 69.30 [52.6 to 78.9] | 53.68 [36.8 to 73.7]
  Change at Week 6 | 2.77 [-5.0 to 6.7] | -2.98 [-16.1 to 8.4] | -3.78 [-16.6 to 16.7] | 4.12 [-8.3 to 22.2]
  Change at Week 14: number analyzed (Participants) | 0 | 0 | 6 | 2
  Change at Week 14 |  |  | -9.90 [-19.4 to 5.0] | 15.55 [3.9 to 27.2]

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of ATYR1940
Time Frame: Cohort 1: Predose, 0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, and 8.0 hours after the start of infusion at Weeks 2 and 5; Cohorts 2 and 3: Predose, 0.5, 1.0, 2.0, 4.0, and 6.0 hours after the start of infusion at Weeks 2, 5, and 13 (Cohort 3 only)
Population: Pharmacokinetic (PK) analysis set included all participants who had baseline samples and sufficient samples collected post-baseline to permit analysis of PK parameters. Here, 'Number Analyzed' signifies participants evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter
Arm/Group | Cohort 1: ATYR1940 0.3 mg/kg | Cohort 2: ATYR1940 1.0 mg/kg | Cohort 3: ATYR1940 3.0 mg/kg
Number analyzed (Participants) | 3 | 6 | 6
nanogram/milliliter
  Week 2 | 1360 (267) | 6800 (752) | 21900 (6960)
  Week 5: number analyzed (Participants) | 3 | 5 | 6
  Week 5 | 1980 (249) | 7490 (1040) | 23800 (8780)
  Week 13: number analyzed (Participants) | 0 | 0 | 5
  Week 13 |  |  | 26200 (14200)

11. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of ATYR1940
Time Frame: as for outcome 10
Population: PK analysis set included all participants who had baseline samples and sufficient samples collected post-baseline to permit analysis of PK parameters. Here, 'Number Analyzed' signifies participants evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1: ATYR1940 0.3 mg/kg | Cohort 2: ATYR1940 1.0 mg/kg | Cohort 3: ATYR1940 3.0 mg/kg
Number analyzed (Participants) | 3 | 6 | 6
hours
  Week 2 | 0.417 (0.144) | 0.500 (0) | 0.500 (0)
  Week 5: number analyzed (Participants) | 3 | 5 | 6
  Week 5 | 0.500 (0) | 0.500 (0) | 0.500 (0)
  Week 13: number analyzed (Participants) | 0 | 0 | 5
  Week 13 |  |  | 0.500 (0)

12. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time 0 to Time t (AUC 0-t) of ATYR1940
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter
Arm/Group | Cohort 1: ATYR1940 0.3 mg/kg | Cohort 2: ATYR1940 1.0 mg/kg | Cohort 3: ATYR1940 3.0 mg/kg
Number analyzed (Participants) | 3 | 6 | 6
nanogram*hour/milliliter
  Week 2 | 5800 (1480) | 24200 (1490) | 82200 (25500)
  Week 5: number analyzed (Participants) | 3 | 5 | 6
  Week 5 | 8550 (1350) | 26500 (2650) | 83700 (25800)
  Week 13: number analyzed (Participants) | 0 | 0 | 5
  Week 13 |  |  | 84400 (36200)

13. Secondary Outcome: Average of Half-life (T1/2) of ATYR1940
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1: ATYR1940 0.3 mg/kg | Cohort 2: ATYR1940 1.0 mg/kg | Cohort 3: ATYR1940 3.0 mg/kg
Number analyzed (Participants) | 3 | 6 | 6
hours
  Week 2 | 3.91 (0.193) | 3.68 (0.354) | 4.33 (0.772)
  Week 5: number analyzed (Participants) | 3 | 5 | 6
  Week 5 | 4.16 (1.04) | 3.91 (1.29) | 4.32 (0.823)
  Week 13: number analyzed (Participants) | 0 | 0 | 5
  Week 13 |  |  | 5.09 (2.64)

ADVERSE EVENTS:
Time Frame: Up to End of Study (up to Week 25)
Description: ITT Analysis Set included all participants who were randomized and received at least 1 dose (full or partial) of study drug.
Arm/Group | Cohort 1: ATYR1940 0.3 mg/kg | Cohort 2: ATYR1940 1.0 mg/kg | Cohort 3: ATYR1940 3.0 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 1/6 | 0/5
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: ATYR1940 0.3 mg/kg (N=3) | Cohort 2: ATYR1940 1.0 mg/kg (N=6) | Cohort 3: ATYR1940 3.0 mg/kg (N=6) | Placebo (N=5)
Infusion-related Reaction (General disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cohort 1: ATYR1940 0.3 mg/kg (N=3) | Cohort 2: ATYR1940 1.0 mg/kg (N=6) | Cohort 3: ATYR1940 3.0 mg/kg (N=6) | Placebo (N=5)
Eyelid Irritation (Eye disorders) | 0 | 1 | 0 | 0
Scintillating Scotoma (Eye disorders) | 0 | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Infusion Site Erythema (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1
Seasonal Allergy (Immune system disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood Pressure Increased (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram PR Shortened (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram QT Prolonged (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram T Wave Inversion (Investigations) | 0 | 1 | 0 | 0
Neutrophil Count Decreased (Investigations) | 0 | 1 | 0 | 0
Protein Urine Present (Investigations) | 0 | 1 | 0 | 0
Pulmonary Function Test Abnormal (Investigations) | 0 | 1 | 0 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 2 | 2
Presyncope (Nervous system disorders) | 0 | 0 | 2 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1
Polymenorrhoea (Reproductive system and breast disorders) | 0/1 | 0/4 | 1/2 | 0/1 — This Adverse event is gender specific.
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 1 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes